CLINICAL TRIAL: NCT01097967
Title: Sleep Disordered Breathing in TIA/Ischemic Stroke: Effects on Short- and Long-term Outcome and CPAP Treatment Efficacy: an Open, Observational, Clinical, Multicentre Trial With a Randomized Arm
Brief Title: Sleep Disordered Breathing in Transient Ischemic Attack (TIA)/Ischemic Stroke and Continuous Positive Airway Pressure (CPAP) Treatment Efficacy
Acronym: SAS-CARE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prof. Claudio Bassetti (Other Government)
Collaborators: Swiss National Science Foundation (Other); Schweizerische Herzstiftung (Other); ResMed (Industry); Philips Respironics (Industry)
Responsible Party: Sponsor-Investigator, Prof. Claudio Bassetti, Dr. med. Claudio Bassetti, Ospedale Civico, Lugano
Organization: Ospedale Civico, Lugano (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EOC.NC.10.01; 320030-125069/1 (Other Grant/Funding Number: Swiss National Science Foundation (SNSF))
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: TIA; Ischemic Stroke
Keywords: Sleep disordered breathing; Continuous Positive Airway Pressure; Sleep apnoea; Markers of atherosclerosis
MeSH Terms: conditions — Ischemic Stroke; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CPAP in sleepy patients with SDB (Active Comparator): SDB defined as AHI >=20 Sleepy defined as Epworth Sleepiness Score >=10
  Interventions: Other: CPAP
- no CPAP in non sleepy patients with SDB (No Intervention): SDB defined as AHI >=20 Sleepy defined as Epworth Sleepiness Score >=10
- CPAP in non sleepy patients with SDB (Active Comparator): SDB defined as AHI >=20 Sleepy defined as Epworth Sleepiness Score >=10
  Interventions: Other: CPAP

INTERVENTIONS:
Other: CPAP
  Arms: CPAP in non sleepy patients with SDB; CPAP in sleepy patients with SDB

SUMMARY:
The study aims to observe the short term effect (3-month) of sleep disordered breathing (SDB) on cardiovascular parameters, heart rate variability, endothelial function and surrogate markers of atherosclerosis after acute cerebrovascular events (ACE). The long-term effect (6-24-month) of Continuous Positive Airway Pressure (CPAP) on clinical vascular outcome, cardiovascular parameters, evolution of surrogate of atherosclerosis heart rate variability and endothelial function after ACE is observed over 24 months. A preventive effect of CPAP therapy on cerebro-vascular events in patients with moderate-severe obstructive SDB without sleepiness after ictus or transient ischaemic attack will be evaluated.

DETAILED DESCRIPTION:
Sleep disordered breathing is an independent risk factor for cardiovascular morbidity and mortality and is frequent in patients with acute cerebrovascular events. In this study the investigators observe the association between sleep disordered breathing, hypertension, stroke and the evolution of blood markers for atherosclerosis as well as the efficacy of Continuous Positive Airway Pressure treatment in patients with acute or subacute cerebrovascular events.

Sleep disordered breathing is an independent risk factor for cardiovascular morbidity and mortality and is frequent in patients with acute cerebrovascular events. In this study the investigators observe the association between sleep disordered breathing, hypertension, stroke and the evolution of blood markers for atherosclerosis as well as the efficacy of Continuous Positive Airway Pressure treatment in patients with acute or subacute cerebrovascular events.

The SAS CARE 1 study is planned to verify whether or not sleep disordered breathing has a detrimental 3 months effect on cardiovascular functions and markers after acute cerebrovascular events. The SAS CARE 2 study is designed to address whether or not the treatment of sleep disordered breathing with CPAP reduces the combined rate of mortality, stroke, cardiovascular events (myocardial infarction/revascularisation/instable angina/ hospitalisation for heart insufficiency) over a 24 months period in patients after acute cerebrovascular events.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 35 years old and < 75 years old
* with clinical diagnosis of TIA or ischemic stroke
* admitted in a Stroke Unit within 2 days from onset of symptoms
* or with TIA or ischemic stroke within the last 60-90 days
* signed Informed Consent

Exclusion Criteria:

* with unstable clinical situation (cardio-respiratory or life-threatening medical conditions)
* currently on CPAP or on CPAP during the last 3 months before stroke
* with non-ischemic events (intracerebral/subarachnoid haemorrhage)
* Patients with coma/stupor
* with borderline obstructive SDB (AHI 10-19)
* with any condition that interferes with the acceptance of CPAP treatment

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2010-07; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Occurence of new vascular events or death in stroke survivors (myocardial infarction, stroke, death) assessed by telephone or reported | 24 monts after stroke
  New vascular events will be assessed by regular telephone interviews at 6,12 and 24 months after stroke

SECONDARY OUTCOMES:
CPAP-Compliance measured by hours of usage | up to 24 months after stroke
  Compliance is monitored for the use of the CPAP by the pulmonary specialist at the patients' routine visits 2-3, 4-6 weeks, 3-6 months, 12 and 24 months after randomisation. The hours ofuse are registered by a chip inserted in the device. Good compliance is, if the device was used > 10 hours per day. Satisfactory compliance is defined for a use of the CPAP for at least 4 hours per night during at least 70% of the nights. Insufficient compliance is defined as < 4 hours per night or less than 70% of nights.
Blood pressure profile (systolic mean, diastolic mean, max, min: general, day, night) measured in mmHg for every patient by ambulatory 24h-BP-devices in the acute stroke phase, after 3 months and after 12 months | up to 12 months after stroke
  Mean systolic and diastolic BP values, minimal and maximum values will be calculated for each patient for each period of time [after stroke: whole measuring period, (36 h) first night, second day, and second night after stroke; 3 months after stroke: whole period (24 h), day, night]. In addition same measurements will be made 12 months after stroke The occurrence of dippers will be registered at baseline (after stroke) and at 3 months. A dipper is defined, if the mean pressure at night is diminished more than 10% (compared to day data). An inverse-dipper is defined if more than 10% augmentation of night pressure will be registered. A deep-deeper is defined the mean pressure at night is diminished more than 20% (compared to day data).
Blood pressure dipping measured by ambulatory 24h-BP-devices in the acute stroke phase, after 3 months and after 12 months | up to 12 months after stroke
  The occurrence of dippers will be registered at baseline (after stroke) and at 3 months and 12 months after stroke. A dipper is defined, if the mean pressure at night is diminished more than 10% (compared to day data). An inverse-dipper is defined if more than 10% augmentation of night pressure will be registered. A deep-deeper is defined the mean pressure at night is diminished more than 20% (compared to day data).

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Bassetti, Professor, Principal Investigator — Universitätsspital Bern (Inselspital) und Universität Bern; Carlo Cereda, Capo CLinica, Study Chair — Neurocentre of Southern Switzerland, Ospedale Civico; Sebastian Ott, MD, Study Chair — Pneumology, University Hospital, Bern; Lino Nobili, Prof. MD, Study Chair — Neurology, Stroke Unit, Ospedale Niguarda, Milan, Italy; Mauro Manconi, MD, Study Chair — Neurocentre of Southern Switzerland, Ospedale Civico; Peter Young, Prof. MD, Study Chair — Universitätsklinik Münster, Zentrum für Schlafmedizin
Locations (5):
- University Hospital Münster, Münster, Germany
- Dipartimento Neuroscienze, Ospedale Niguarda, Milan, Lombardy, Italy
- Switzerland (3):
  - Inselspital, Universitätsklinik für Pneumologie, Bern, Canton of Bern
  - Ospedale San Giovanni, Bellinzona, Canton Ticino
  - Neurocenter of Southern Switzerland, Ospedale Civico, Lugano, Canton Ticino

REFERENCES:
- [Background] Bassetti C, Aldrich MS, Chervin RD, Quint D. Sleep apnea in patients with transient ischemic attack and stroke: a prospective study of 59 patients. Neurology. 1996 Nov;47(5):1167-73. doi: 10.1212/wnl.47.5.1167. PMID 8909424
- [Background] Bassetti C, Aldrich MS. Sleep apnea in acute cerebrovascular diseases: final report on 128 patients. Sleep. 1999 Mar 15;22(2):217-23. doi: 10.1093/sleep/22.2.217. PMID 10201066
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Bassetti CL, Milanova M, Gugger M. Sleep-disordered breathing and acute ischemic stroke: diagnosis, risk factors, treatment, evolution, and long-term clinical outcome. Stroke. 2006 Apr;37(4):967-72. doi: 10.1161/01.STR.0000208215.49243.c3. Epub 2006 Mar 16. PMID 16543515
- [Background] Martinez-Garcia MA, Soler-Cataluna JJ, Ejarque-Martinez L, Soriano Y, Roman-Sanchez P, Illa FB, Canal JM, Duran-Cantolla J. Continuous positive airway pressure treatment reduces mortality in patients with ischemic stroke and obstructive sleep apnea: a 5-year follow-up study. Am J Respir Crit Care Med. 2009 Jul 1;180(1):36-41. doi: 10.1164/rccm.200808-1341OC. Epub 2009 Apr 30. PMID 19406983
- [Derived] Pace M, Camilo MR, Seiler A, Duss SB, Mathis J, Manconi M, Bassetti CL. Rapid eye movements sleep as a predictor of functional outcome after stroke: a translational study. Sleep. 2018 Oct 1;41(10). doi: 10.1093/sleep/zsy138. PMID 30032306
- [Derived] Manconi M, Zavalko I, Cereda C, Pisarenco I, Ott S, Fulda S, Bassetti CL. Longitudinal polysomnographic assessment from acute to subacute phase in infratentorial versus supratentorial stroke. Cerebrovasc Dis. 2014;37(2):85-93. doi: 10.1159/000356323. Epub 2014 Jan 16. PMID 24435018
- [Derived] Cereda CW, Petrini L, Azzola A, Ciccone A, Fischer U, Gallino A, Gyorik S, Gugger M, Mattis J, Lavie L, Limoni C, Nobili L, Manconi M, Ott S, Pons M, Bassetti CL. Sleep-disordered breathing in acute ischemic stroke and transient ischemic attack: effects on short- and long-term outcome and efficacy of treatment with continuous positive airways pressure--rationale and design of the SAS CARE study. Int J Stroke. 2012 Oct;7(7):597-603. doi: 10.1111/j.1747-4949.2012.00836.x. Epub 2012 Jul 19. PMID 22812731
- See also: Click here to see more information about our hospital — http://www.eoc.ch
- See also: provides financial support for the study — http://www.swissheart.ch